CLINICAL TRIAL: NCT06361719
Title: Efficacy of a Ready to Feed (RTF) Starter Liquid Infant Formula Containing 2'FL and LNnT in Chinese Infants: A Double-blind, Randomized Controlled Trial Including a Breastfed Reference Group
Brief Title: Efficacy of Two HMOs in Chinese Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2312INF
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy Infants
Keywords: Human Milk Oligosaccharides; Infant gut microbiota; Infant gut health; Immune response; Growth; Tolerance
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (EG) (Experimental): Starter infant formula supplemented with two HMOs. Following the intervention period, the infants will consume a standard infant follow-up formula (non-trial formula).
  Interventions: Other: Experimental Group (EG)
- Control Group (CG) (Active Comparator): Starter infant formula not supplemented with two HMOs. Following the intervention period, the infants will consume a standard infant follow-up formula (non-trial formula).
  Interventions: Other: Control Group (CG)
- Breastfed Group (BG) (No Intervention): Breast Milk

INTERVENTIONS:
Other: Experimental Group (EG) — Starter infant formula will be administered to the participants orally, ad libtium to 6 months, after which they will transfer to a classical follow-up formula (non-trial formula) until the end of the trial (12 months of age).
  Arms: Experimental Group (EG)
Other: Control Group (CG) — Starter infant formula will be administered to the participants orally, ad libtium to 6 months, after which they will transfer to a classical follow-up formula (non-trial formula) until the end of the trial (12 months of age).
  Arms: Control Group (CG)

SUMMARY:
This is a randomized, controlled, double-blind, intervention trial of healthy male and female term infants to evaluate the efficacy of the 2 HMOs on beneficially modulating the gut microbiota, gut maturation, gut barrier integrity, immune response, and other developmental outcomes in healthy Chinese infants. The trial consists of 2 randomized formula-fed groups, and a non-randomized breastfed reference group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female infants of post-natal age of 3-14 days (date of birth = day 0), inclusive, at enrolment
* Evidence of personally signed and dated informed consent document indicating that the infant's parent(s)/ legally accepted representatives LAR have been informed of all pertinent aspects of the trial.
* Infants whose parent(s) have reached the legal age of majority in China.
* Infants whose parent(s)/LAR are willing and able to comply with scheduled visits, and the requirements of the trial protocol.
* Infants whose parent(s)/LAR can be contacted directly by telephone throughout the trial.
* Infants whose parent(s)/LAR have a working freezer.
* Singleton, healthy, full-term gestational birth (≥ 37 completed weeks of gestation), with a birth weight of ≥ 2.5 kg and ≤ 4.5 kg.
* For the formula-fed groups: infant is exclusively consuming and tolerating a cow' s milk infant formula for at least 3 days prior to enrolment. The infant's mother has independently elected not to breastfeed.
* For the breastfed reference group: infant has been exclusively consuming breastmilk since birth (small amounts of other feedings allowed during the first three days of life before breastfeeding is well-established) and the infant's mother has made the decision to continue exclusively breastfeeding until at least 3 months of age.

Exclusion Criteria:

* Infants with conditions requiring infant feedings other than those specified in the protocol.
* Infants receiving complementary foods or liquids defined as 4 or more teaspoons per day or approximately 20 g per day of complementary foods or liquids at or prior to enrolment.
* Infants who have a medical condition or history that could increase the risk associated with trial participation or interfere with the interpretation of trial results, including: Evidence of major congenital malformations (e.g., cleft palate, extremity malformation). Documented or suspected systemic or congenital infections (e.g., human immunodeficiency virus, cytomegalovirus, syphilis). Previous or ongoing severe medical or laboratory abnormality (acute or chronic) which, in the judgment of the investigator, would make the infant inappropriate for entry into the trial.
* Infants who are presently receiving or have received prior to enrolment probiotic supplements or any of the following: medication(s) or supplement(s) which are known or suspected to affect the following: fat digestion, absorption, and/or metabolism (e.g., pancreatic enzymes); stool characteristics and microbiota (e.g., oral and systemic antibiotics, glycerine suppositories, bismuth-containing medications, docusate, Maltsupex, or lactulose); growth (e.g. insulin or growth hormone); gastric acid secretion.
* Currently participating or having participated in another clinical trial since birth.
* Infant who has known or suspected cows' milk protein intolerance / allergy, lactose intolerance, soy intolerance / allergy.

Ages: 3 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 262 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Bifidobacteria abundance in fecal samples | just prior to 3 months of age
  Bifidobacteria abundance using qPCR technology

SECONDARY OUTCOMES:
Gut microbiota composition | From enrollment until 12 months of age
  Relative abundance of beneficial and potentially pathogenic species using next generation sequencing (NGS) technology
Fecal metabolism | From enrollment until 12 months of age
  Fecal pH analyzed using HPLC as well as targeted or untargeted metabolomics profiling
Fecal metabolism | From enrollment until 12 months of age
  Short chain fatty acids analyzed using HPLC as well as targeted or untargeted metabolomics profiling
Fecal markers of intestinal immune health | From enrollment until 6 months of age
  Fecal secretory IgA measured by ELISA
Fecal markers of gut barrier function | From enrollment until 6 months of age
  Calprotectin measured by ELISA
Fecal markers of gut barrier function | From enrollment until 6 months of age
  α-1-antitrypsin measured by ELISA
Fecal markers of gut barrier function | From enrollment until 6 months of age
  Lipocalin-2 measured by ELISA
Fecal markers of inflammation | From enrollment until 6 months of age
  Levels of cytokines such as IL-1β measured by ELISA
Fecal markers of inflammation | From enrollment until 6 months of age
  Levels of cytokines such as IFN-γ measured by ELISA
Fecal markers of inflammation | From enrollment until 6 months of age
  Levels of cytokines such as TNF-α measured by ELISA
Stool patterns | From enrollment until 14 days
  Stool frequency, consistency, and difficulty in passing stools assessed using a 1-day retrospective stool consistency diary (24-hr recall)
Stool patterns | From enrollment until 12 months of age
  Stool frequency, consistency, and difficulty in passing stools assessed using a 3-day prospective collection recorded in the stool consistency diary.
GI symptoms and behaviors | From enrollment until 6 months of age
  IGSQ-13 Questionnaire
Immune competence | From enrollment until 12 months of age
  Pediatric Immune System Index score
Infant sleep duration and night-time wakings per 24 hours | From enrollment until 6 months of age
  Brief infant sleep questionnaire (BISQ)
Infant Health Related Quality of Life | From enrollment until 6 months of age
  Infant Toddler Quality of Life Questionnaire (ITQoL -SF47)
Growth | From enrollment until 12 months of age
  Weight (g) and corresponding Z-scores
Growth | From enrollment until 12 months of age
  Length (cm) and corresponding Z-scores
Growth | From enrollment until 12 months of age
  Head circumference (cm) and corresponding Z-scores
Growth | From enrollment until 12 months of age
  Weight gain and corresponding Z-scores
Growth | From enrollment until 12 months of age
  Length gain, corresponding Z-scores
Physical Examination | At enrollment and at 12 months of age
Infant Illness | From enrollment until 12 months of age
  Infant Illness Diary
Infant illness, infections and medication usage | From the time the informed consent form has been signed at enrollment infant age less than 3 days until 12 months of age
  AEs and Serious Adverse Events (SAEs)
Medication use (type and duration) | From enrollment until 12 months of age
  Concomitant medication form and Infant Illness Diary

OTHER OUTCOMES:
Formula feeding | From enrollment until 12 months of age
  Total quantity of milk consumed for formula-feeding
Breastfeeding | From enrollment until 12 months of age
  The frequency of breastfeeding, duration and type of breastfeeding (exclusive, predominant, partial)
Infant dietary pattern | From 6 months of age until 12 months of age
  3-day food diary

CONTACTS AND LOCATIONS:
Overall Officials: Wei Cai, MD, Principal Investigator — Shanghai Institute for Pediatric Research, Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- The International Peace Maternity & Child Health Hospital of China Welfare Institute, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Y, Le Roy CI, Li J, Han S, Liu Z, Lahiry A, Sahu H, Li Q, Dong J, Mondragon A, Samuel TM, Cai W. Efficacy of a Ready-to-Feed Starter Liquid Infant Formula Containing 2-Fucosyllactose and Lacto-N-Neotetraose in Chinese Infants: Protocol for a Double Blind, Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 31;14:e66489. doi: 10.2196/66489. PMID 41172301